CLINICAL TRIAL: NCT02679378
Title: Clinical Study of the ClearSight™ System to Evaluate the Ability to Distinguish Malignant From Non-malignant Breast Tissue by Comparing MR Measurements of Freshly Excised Breast Tissue to Histopathology
Brief Title: Exploratory Study Comparing ClearSight System 2D Map to Post Surgery Histopathological Analysis in Lumpectomy
Status: Completed | Type: Observational
Sponsor: Clear Cut Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 710CLD Rev. 02
Record Dates: First submitted 2016-01-25; First posted 2016-02-10 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ClearSight™ System: To assess the ability of the ClearSight™ System to detect malignant tissue less than or equal to 1 mm of margins of excised breast specimen in breast conserving surgery when compared to histopathological assessment.
  Interventions: Device: ClearSight™ System

INTERVENTIONS:
Device: ClearSight™ System — comparing ClearSight system to histopathological to determine negative-margins in breast conserving surgery.

SUMMARY:
Prospective, single-arm, multicenter, open label, non-randomized exploratory clinical study comparing ClearSight system to histopathological to determine negative-margins in breast conserving surgery.

DETAILED DESCRIPTION:
This study is a multicenter, non-randomized, cross-sectional comparative exploratory study comparing the ClearSight System 2D map results to post surgery histopathological analysis of excised mass in lumpectomy surgery. The Efficacy Objective is to assess the ability of the ClearSight™ System to detect malignant tissue less than or equal to 1 mm of margins of excised breast specimen in breast conserving surgery using histopathological assessment as reference. The Safety Objective is that all adverse events, serious adverse events (SAE) will be reported according to local regulations. The actual reporting is discussed in section 0. No device-related adverse events are expected. For more information please refer to the Investigator Brochure.

ELIGIBILITY:
Inclusion Criteria:

1. Women histologically diagnosed with carcinoma of the breast, scheduled for primary lumpectomy (partial mastectomy) procedure.
2. Age ≥18.
3. Signed ICF

Exclusion Criteria:

1. Prior surgical procedure in the same breast within 12 months prior to the surgery date.
2. Recurrent breast cancer surgery.
3. Neoadjuvant chemotherapy.
4. Previous radiation therapy to the operated breast.
5. Pregnant / breast feeding.
6. Participating in any other study that might affect results.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — WOMEN
Study Population: Patients diagnosed with primary breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Malignant and non-malignant breast tissues will be assessed by ClearSight™ to detect malignant tissue less than or equal to 1 mm of margins of excised breast specimen in breast conserving surgery using histopathological assessment as reference | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christine B. Teal, Dr., Principal Investigator — The George Washington University (GWU)
Locations (5):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - The George Washington University Hospital (GWU), Washington D.C., District of Columbia
- Israel (3):
  - Kaplan Medical Center, Rehovot
  - Assuta Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin

IPD SHARING:
Plan to Share IPD: Undecided